CLINICAL TRIAL: NCT02332330
Title: A Post-market Prospective Study of the VGS VEST (Venous External Support), Supporting Saphenous Vein Grafts for Coronary Bypass Graft Surgery in Patients With Severe Coronary Heart Disease
Brief Title: CD0104 VEST II Post Marketing Surveillance Study
Acronym: VEST II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Graft Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD0104
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Bypass Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VEST (Experimental)
  Interventions: Device: VEST

INTERVENTIONS:
Device: VEST

SUMMARY:
This study is designed to collect post market data on use of the VEST, particularly on saphenous vein grafts to the right territory of the heart.

DETAILED DESCRIPTION:
The primary objective is to test the early-mid term patency rate of VEST supported Right Coronary Artery (RCA) bypass grafts. The research participants will undergo CABG preparations and CABG procedure routinely as is the standard of care. During the procedure the VEST will be implanted on the vein graft to the Right Coronary Artery according to the IFU. Perioperative care is according to standard of care. Upon discharge patient will be prescribed statins and aspirin for 6 months. Patient will attend a routine clinic visit 4-6 weeks post operatively. The last study visit will occur 3-6 months post operatively. Patients will undergo a noninvasive coronary CT angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for on-pump CABG on clinical grounds
2. At least one vein graft bypass indicated for right coronary artery and LIMA indicated for the LAD on clinical grounds
3. Appropriately sized and accessible target coronary arteries, with a minimum diameter of 1.5 mm and adequate vascular bed, as assessed from the pre-operative cardiac angiography.

Exclusion Criteria:

1. Concomitant non-CABG cardiac procedure
2. Prior cardiac surgery
3. Emergency CABG surgery (cardiogenic shock, inotropic pressure support, IABP)
4. Contraindication for on-pump CABG with cardioplegic arrest (e.g. severely calcified aorta)
5. Calcification at the intended anastomotic sites, as assessed upon opening of the chest and before VEST implantation.
6. Prior debilitating stroke less than 1 year before surgery
7. Severe renal dysfunction (Cr>2.0 mg/dL)
8. Concomitant life-threatening disease likely to limit life expectancy to less than 2 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Vein graft patency by CT angiography | 3-6 monthws
MACCE | 3-6 months
  Major adverse cardiac and cerebral events

CONTACTS AND LOCATIONS:
Overall Officials: David P Taggart, Professor, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (2):
- Krankenhaus der Barmherzigen Bruder, Trier, Germany
- The John Radcliffe Hospital, Oxford, United Kingdom